CLINICAL TRIAL: NCT07241754
Title: Predictors of Anti-seizure Medication Resistance in Pediatric Epilepsy
Brief Title: Predictors of Drug Resistant Epilepsy Among Pediatric Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dalia Abdelrahim Fakhry Hussein, Principal Investigator, Assiut University
Other Study IDs: Drugs resistant epilepsy
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Epilepsy; Seizure; Resistance
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. This study aims to determine the main predictors of drug resistance in pediatric epilepsy by examining clinical data, EEG abnormalities, and neuroimaging results, in order to support early identification of resistant cases and improve treatment strategies .
2. Early introduction of new lines of treatment in case of refractory epilepsy as : Ketogenic diet , Rituximab and solumedrol

DETAILED DESCRIPTION:
Epilepsy is among the most prevalent chronic neurological disorders in the pediatric population, affecting approximately 0.5-1% of children worldwide . It is characterized by recurrent, unprovoked seizures resulting from abnormal, excessive, or synchronous neuronal activity in the brain. Epilepsy in childhood represents a major public health concern, not only because of its relatively high incidence, but also due to its significant impact on neurodevelopment, cognitive functions, psychosocial well-being, and overall quality of life .

Despite the remarkable advances in pharmacological therapy, the cornerstone of epilepsy management remains antiseizure medications (ASMs). More than two-thirds of children with epilepsy achieve satisfactory seizure control with one or two appropriately chosen medications. However, a considerable proportion-estimated at 20-40%-develop drug-resistant epilepsy (DRE) . According to the International League Against Epilepsy (ILAE), DRE is defined as the failure to achieve sustained seizure freedom after adequate trials of at least two well-tolerated and appropriately selected ASMs, whether administered as monotherapy or in combination . Children with DRE are at a particularly high risk of poor neurocognitive outcomes, behavioral problems, injury, psychosocial difficulties, and even increased mortality .

Given the serious consequences of uncontrolled epilepsy, early identification of patients at risk for ASM resistance is of paramount importance. Predictors of drug resistance in pediatric epilepsy have been widely studied, although results vary across different populations and study designs. Factors frequently reported include early age at seizure onset, high initial seizure frequency, abnormal developmental history, specific electroencephalographic (EEG) abnormalities, structural brain lesions, identifiable genetic syndromes, and poor response to the first-line ASM . Recognition of these predictors can enable clinicians to stratify patients into risk categories, anticipate treatment challenges, and implement timely alternative interventions such as epilepsy surgery, ketogenic diet, or neuromodulation .

Moreover, exploring predictors of ASM resistance in children is not only clinically relevant, but also contributes to a better understanding of the pathophysiology of epilepsy and its heterogeneous nature. By delineating the factors that influence treatment outcomes, researchers and clinicians may be able to develop more targeted therapeutic strategies, improve prognostic counseling for families, and ultimately enhance the overall management of pediatric epilepsy .

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-18 years with a confirmed diagnosis of epilepsy.
* Both males and females will be included.

Exclusion Criteria:

* Children younger than 1 year or older than 18 years.
* Patients with acute symptomatic seizures (e.g., febrile seizures, metabolic or infectious causes) or pseudo refractory epilepsy (e .g. syncope or uncorrect ASMs)
* Patients controlled on antiseizure medications
* Refusal of parents or guardians to participate in the study

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will include children and adolescents aged 1 month to 18 years with a confirmed diagnosis of epilepsy according to ILAE criteria, who are followed at pediatric neurology clinics and epilepsy units. Eligible participants must have received antiepileptic drug therapy for at least 6 months and have available clinical records, EEG findings, and neuroimaging results. Patients with only acute symptomatic seizures, progressive neurodegenerative diseases, prior epilepsy surgery, or incomplete data will be excluded. Participants will be recruited consecutively from outpatient and inpatient services, with informed consent obtained from caregivers and assent from older children when appropriate.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2026-12-29 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Predictors of Drug Resistance in Pediatric Epilepsy | through 12 months of follow-up.
  Identification of clinical, EEG, and neuroimaging predictors of resistance to anti-seizure medications in pediatric epilepsy, to enable early recognition and guide treatment strategies.

SECONDARY OUTCOMES:
Assessed from the time of diagnosis of drug resistance up to 12 months following initiation of the alternative treatment. | Assessed from the time of diagnosis of drug resistance up to 6 to 12 months following initiation of the alternative treatment.
  Evaluation of the role of introducing alternative treatment modalities (such as ketogenic diet, rituximab, and solumedrol) in pediatric patients who develop refractory epilepsy, and their impact on seizure control and clinical outcomes.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Loscher W, Potschka H, Sisodiya SM, Vezzani A. Drug Resistance in Epilepsy: Clinical Impact, Potential Mechanisms, and New Innovative Treatment Options. Pharmacol Rev. 2020 Jul;72(3):606-638. doi: 10.1124/pr.120.019539. PMID 32540959
- [Result] Devinsky O, Vezzani A, O'Brien TJ, Jette N, Scheffer IE, de Curtis M, Perucca P. Epilepsy. Nat Rev Dis Primers. 2018 May 3;4:18024. doi: 10.1038/nrdp.2018.24. PMID 29722352
- [Result] Sillanpaa M, Schmidt D. Natural history of treated childhood-onset epilepsy: prospective, long-term population-based study. Brain. 2006 Mar;129(Pt 3):617-24. doi: 10.1093/brain/awh726. Epub 2006 Jan 9. PMID 16401617
- [Result] Kwan P, Brodie MJ. Early identification of refractory epilepsy. N Engl J Med. 2000 Feb 3;342(5):314-9. doi: 10.1056/NEJM200002033420503. PMID 10660394
- [Result] Aaberg KM, Gunnes N, Bakken IJ, Lund Soraas C, Berntsen A, Magnus P, Lossius MI, Stoltenberg C, Chin R, Suren P. Incidence and Prevalence of Childhood Epilepsy: A Nationwide Cohort Study. Pediatrics. 2017 May;139(5):e20163908. doi: 10.1542/peds.2016-3908. Epub 2017 Apr 5. PMID 28557750
- [Result] Russ SA, Larson K, Halfon N. A national profile of childhood epilepsy and seizure disorder. Pediatrics. 2012 Feb;129(2):256-64. doi: 10.1542/peds.2010-1371. Epub 2012 Jan 23. PMID 22271699